CLINICAL TRIAL: NCT05904730
Title: Phase I Clinical Trials Investigating the Potential Efficacy of Axitinib in Patients With a BRCA 1/2 Mutations Independent of HER2 Expression With Progression After Previous Treatment
Brief Title: Phase I Clinical Trials Investigating the Potential Efficacy of Axitinib in Patients With a BRCA 1/2 Mutations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lynkcell Europe (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6334536
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer; Ovarian Cancer; Breast Neoplasms; Ovarian Neoplasms; BRCA Mutation; HER2-positive Breast Cancer; HER2-negative Breast Cancer; HER-2 Protein Overexpression
Keywords: Axitinib; Inlyta; AG-013736
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms | interventions — Axitinib

STUDY DESIGN:
Intervention Model Description: The starting dose of Axitinib is 5 mg BID administered orally with food.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Axitinib is 5 mg BID administered orally (Experimental): The starting dose of Axitinib 5 mg BID administered orally with food.
  Interventions: Drug: Axitinib

INTERVENTIONS:
Drug: Axitinib — The starting dose of axitinib is 5 mg twice daily by mouth with meals. (reception is desirable at the same time every day)
  Other Names: AG-013736; INLYTA

SUMMARY:
This Clinical Trial is investigating the potential efficacy of axitinib after genetic testing in BRCA 1/2 Mutation patients, regardless of HER2 expression, who have progressed after at least one line of standard treatment or for whom there is no consensus treatment approach.

The use of Axitinib may help physicians plan for more effective patient care in combination with existing treatment protocols.

DETAILED DESCRIPTION:
This Clinical Trial is investigating the potential efficacy of axitinib after genetic testing in BRCA 1/2 Mutation patients, regardless of HER2 expression, who have progressed after at least one line of standard treatment or for whom there is no consensus treatment approach.

The use of Axitinib may help physicians plan for more effective patient care in combination with existing treatment protocols.

The addition of Axitinib to existing treatment protocols and to fractionated irradiation without functional normalization of the tumor vasculature can significantly improve response to therapy, contributing to the breakdown of the metabolic symbiosis of adaptive drug resistance.

ELIGIBILITY:
Inclusion Criteria:

* histologically and immunohistochemically confirmed status of the tumor process
* мale or female, age ≥ 18 years
* Karnofsky performance status ≥ 60
* signed informed consent and willingness/ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures

Exclusion Criteria:

* Grade 3 bleeding NCI CTCAE prior to study enrollment
* cardiac arrhythmias ≥2 according to NCI CTCAE with a corrected QT interval (QTcF) on the screening ECG >480 ms.
* pregnancy or breastfeeding. All female subjects of reproductive potential must have a negative pregnancy test (serum) prior to enrollment. Male subjects must be surgically sterile or must consent to the use of effective contraception during therapy.
* severe acute or chronic psychiatric condition or disorder with risk associated with participation in the study
* congestive heart failure (CHF) class III or higher according to the New York Heart Association (NYHA)
* subjects with arterial thrombotic events / venous thrombosis in the previous 12 months (axitinib has never been studied in this population)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-07-11 (Actual); Primary Completion 2024-11-09 (Actual); Study Completion 2024-12-26 (Actual)

PRIMARY OUTCOMES:
Antitumor effect of axitinib (INLYTA) among patients with solid tumors with BRCA 1/2 mutations independent of HER2 expression, with progression after previous treatment, including radiotherapy | up to 90 days
  Percent reduction of longest diameter of tumor and (or) metastases in millimeters

CONTACTS AND LOCATIONS:
Locations (2):
- Ukraine (2):
  - Trials TEAM, Dnipro
  - Trials TEAM, Kyiv

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/24755544/
- See also: Related Info — https://hccpjournal.biomedcentral.com/articles/10.1186/s13053-021-00193-y